CLINICAL TRIAL: NCT03874247
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, Multi-center Phase III Clinical Trial to Evaluate the Efficacy and Safety of 'Pelubiprofen Controlled Released Tab.' in Acute Traumatic Injury
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of 'Pelubiprofen Controlled Released Tab.' in Acute Traumatic Injury
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW9801-302
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Acute Traumatic Injury
MeSH Terms: interventions — pelubiprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelubiprofen (Experimental)
  Interventions: Drug: pelubiprofen 45mg
- Pelubiprofen placebo (Placebo Comparator)
  Interventions: Drug: pelubiprofen placebo

INTERVENTIONS:
Drug: pelubiprofen 45mg — bid for 3 days after meal
  Arms: Pelubiprofen
Drug: pelubiprofen placebo — bid for 3 days after meal
  Arms: Pelubiprofen placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel, multi-center phase III clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, ages over 19 years
* Patients with post traumatic acute pain within 48 hr(sprain/strain)
* Patient whose pain scale is over 50 mm(VAS score)

Exclusion Criteria:

* Patients with chronic pain
* Presence of a fracture or more than one injury
* Previous adverse reaction or known allergy to NSAIDs

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
SPID-D3 | Day 3
  Sum of Pain Intensity Differences(100 mm pain VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea